CLINICAL TRIAL: NCT01864512
Title: A Prospective, Multicenter Study on the Alteration of Different Immune Parameters in ITP Patients Receiving Eltrombopag Treatment.
Brief Title: Alteration of Different Immune Parameters in Immune Thrombocytopenia （ITP） Patients Receiving Eltrombopag Treatment
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ming Hou, professor, Shandong University
Other Study IDs: ITP-eltrombopag
Record Dates: First submitted 2013-05-17; First posted 2013-05-29 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-06

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; eltrombopag; immune regulation
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens were retained for PCR, western blotting and FACS analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ITP patients receiving eltrombopag therapy

SUMMARY:
This project was undertaken by Qilu Hospital of Shandong University and other well-known hospitals in China. In order to report the alteration of Different Immune Parameters in ITP Patients Receiving Eltrombopag Treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy of oral eltrombopag as a thrombopoietic agent treating previously treated chronic Chinese ITP patients and investigate the alteration of Different Immune Parameters after eltrombopag therapy.

Approximately 30 eligible subjects with primary ITP who have not responded to or have relapsed after previous treatment for ITP will be selected. The initial dose of eltrombopag administration is 25 mg orally once daily. During the 6 weeks follow-up, dose of investigational product will be adjusted according to the weekly subject platelet count, and a battery of immune parameters will be monitored at the end of each week. Additionally, the efficacy of oral eltrombopag for ITP will be assessed after 6 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old.
2. Diagnosed with ITP for at least 12 months prior to screening, and have a platelet count of <30 X109/L on Day 1 (or within 48 hours prior to dosing on Day 1).
3. Patients who have no response or relapsed after splenectomy. Or patients who have not been splenectomised and have either not responded to one or more prior therapies (except splenectomy), or who have relapsed prior therapy.
4. Previous therapy for ITP including rescue must have been completed at least 2 weeks prior to randomization, and other TPO-R agonists, such as romiplostim or recombinant human thrombopoietin (rhTPO), must have been completed for more than 30 days before enrollment.
5. Subjects treated with maintenance immunosuppressive therapy must be receiving a dose that has been stable for at least 1 month.
6. No pre-existing cardiac disease within the last 3 months. No arrhythmia known to increase the risk of thrombolic events (e.g. atrial fibrillation), or patients with a Corrected QT interval (QTc) >450msec or QTc >480 for patients with a Bundle Branch Block.
7. No history of clotting disorder, other than ITP.
8. A complete blood count (CBC), within the reference range, with the following exceptions:

   * Platelets <30×109/L on Day 1 (or within 48hours of Day 1) is required for inclusion,
   * Hemoglobin: females and males 10.0 g/dl are eligible for inclusion,
   * Absolute neutrophil count (ANC) ≥1500/µL (1.5×109/L) is required for inclusion
9. Blood chemistry test result no exceed normal by more than 20%. Total albumin must not be below the lower limit of normal (LLN) by more than 10%.
10. Subject is non-childbearing potential of childbearing potential and use acceptable methods of contraception from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study.

    -

Exclusion Criteria:

1. Patients with any prior history of arterial or venous thrombosis, AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, antiphospholipid syndrome, etc).
2. Any clinically relevant abnormality, other than ITP,which in the opinion of the investigator makes the subject unsuitable for participation in the study.
3. Female subjects who are nursing or pregnant at screening or pre-dose on Day 1.
4. History of alcohol/drug abuse or dependence within 12 months of the study.
5. Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
6. Subjects who have previously received eltrombopag therapy.
7. Subject has consumed aspirin, aspirin-containing compounds, salicylates, anticoagulants, quinine or non-steroidal anti-inflammatories (NSAIDs) for >3 consecutive days within 2 weeks of the study start and until the end of the study.
8. Consumption of any herbal or dietary supplements, excluding vitamin or mineral supplements, within 1 week of the study start.
9. History of platelet aggregation that prevents reliable measurement of platelet counts.
10. An abnormality in bone marrow examination result, other than ITP, identified on the screening examination, which in the opinion of the investigator makes the subject unsuitable for participation in the study.
11. Any laboratory or clinical evidence for HIV infection; any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subject screening. Laboratory test at screening show evidence for hepatitis C infection or hepatitis B infection.
12. Patients expected to require rescue on Day 1 of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese chronic primary immune thrombocytopenia (ITP) adult subjects who have not responded to or have relapsed after previous treatment for ITP, including first line therapy and /or splenectomy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 6 weeks
  1. Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  2. Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  3. No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
Alteration of Different Immune Parameters | 6 weeks
  immune parameters,including expression of CD14,FcgammaRI,FcgammaRIIa/IIb and FcgammaRIII on monocyte/macrophages, will be determined once weekly till the end of the sixth week.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Peng, Doctor, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu XG, Liu S, Feng Q, Liu XN, Li GS, Sheng Z, Chen P, Liu Y, Wei Y, Dong XY, Qin P, Gao C, Ma C, Zhang L, Hou M, Peng J. Thrombopoietin receptor agonists shift the balance of Fcgamma receptors toward inhibitory receptor IIb on monocytes in ITP. Blood. 2016 Aug 11;128(6):852-61. doi: 10.1182/blood-2016-01-690727. Epub 2016 Jun 8. PMID 27281793